CLINICAL TRIAL: NCT03899584
Title: Quality of Life, Efficacy and Safety of High Doses of 4-aminopyridine in Patients With Clinically Complete Chronic Spinal Cord Injury: Multicenter, Randomized, Double Blind, Placebo Controlled Clinical Trial
Brief Title: High Doses of 4-aminopyridine in Clinically Complete Chronic Spinal Cord Injury Patients.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-785-073
Record Dates: First submitted 2019-02-13; First posted 2019-04-02 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injuries; Chronic
Keywords: 4-Aminopyridine; erectile function; tetraplegia; rehabilitation; questionnaires; paraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Bronchiolitis Obliterans Syndrome; Quadriplegia; Paraplegia | interventions — 4-Aminopyridine; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with 4-aminopyridine (Active Comparator): The 4-aminopyridine will be administered in the form of gelatin capsules containing 4-aminopyridine 10 mg and microcrystalline cellulose as excipient. The dose of 4-aminopyridine will increase 10 mg / every 2 to 4 weeks until reaching the maximum dose proposed by weight ( maximum 1 mg / kg / d).
  Interventions: Drug: 4-Aminopyridine
- Placebo oral capsule (Placebo Comparator): Patients randomized to the placebo sequence will receive placebo in the same way as those who will take 4-AP. They will be blinded to the fact that they are taking placebo and the capsules will be identical in appearance to the intervention capsules.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: 4-Aminopyridine — Each patient will take 10 mg per kilogram of weight (example: a person weighing 60 kg, will take two capsules three times a day after meals, for a total of 6 capsules / day). Each capsule will contain 10 milligrams of 4-Aminopyridine that will allow to be administered sequentially at progressively higher doses / day. The dose of 4-aminopyridine will increase 10 mg / 2 to 4 weeks.
  Other Names: 4-AP
  Arms: Treatment with 4-aminopyridine
Drug: Placebo oral capsule — The placebo arm will include a placebo of microcrystalline cellulose.
  Other Names: Microcrystalline cellulose
  Arms: Placebo oral capsule

SUMMARY:
150 patients with clinically complete chronic spinal cord Injury will be included in a randomized, parallel, placebo controlled, multi-centric, phase III trial. Patients will be evaluated before starting the medication, and at the end of the treatment in the locomotor, sensory, grade of independence, sensitivity and control of bladder and anal sphincters, quality of life, and psychogenic erection in males. Patients will be divided randomly into two groups where one will receive placebo and the other one 4-Aminopyridine (4-AP) in a maximum of 30 weeks in increasing doses.

DETAILED DESCRIPTION:
Consecutive patients with chronic AIS A tetraplegic or paraplegic with an MRI showing cord continuity will be recruited in the departments of neurology, neurosurgery or rehabilitation from hospitals of Social Security Mexican Institute (IMSS) in 8 states . Just patients who meeting inclusion criteria, will be selected for the study until reach 150. After signing an informed consent, they will be randomized into 75 for the intervention arm and 75 for the placebo arm. All patients will receive capsules for daily consumption according to their assignment. They will receive ascending doses of the drug starting with 10 milligrams and progressively increasing every 2 to 4 weeks 10 mg until reaching the maximum dose proposed according to weight (maximum 1 mg/kg/d). Questionnaires and functional evaluations will be administered at the beginning of the study, and at the end of the treatment to evaluate the efficacy. The evaluations include the International Standards for Neurological Classification of Spinal Cord Injury motor and sensory Scale, the Spinal Cord Injury Independence Measure (SCIM III), quality of life (SF-36), sphincter bladder/anal sensation/control in both genders and psychogenic erection in males as primary outcomes.

After the follow-up period, all test results will be analyzed and compared to determine the efficacy and safety of 4-aminopyridine. The Mann-Whitney U and Chi-square test will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria: Patients with spinal cord injury (SCI) will be eligible for the study if they meet the following criteria:

1. Chronic AIS A tetraplegia or paraplegia for more tan 2 years before the study begin.
2. MRI showing cord continuity.
3. Neurologic Injury level of C4-T12.
4. Medically stable and able to breathe independently.
5. Stable neurologic deficits for more than 60 days before the study.
6. The absence of antiepileptic antecedent and electroencephalogram without epileptic activity.
7. They have maintained some type of rehabilitation after injury in the affected limbs and paralyzed extremities without passive limitations (healthy joints)
8. For females: postmenopausal or surgically sterile, or using an acceptable method of birth control.

Exclusion Criteria:

1. Pressure ulcers, skin infections, or phlebitis
2. History of cardiovascular disease (syncope, arrhythmia, or myocardial infarction within the last two years), systolic blood pressure greater than 150 or less than 70 mm Hg, diastolic blood pressure greater than 110 or less than 50 mm Hg, or heart rate greater than 110 or less than 50 beats/minute; impaired hepatic function (total hepatic enzyme or bilirubin levels greater than 2 times the upper limits of normal) or impaired renal function (creatinine level greater than 2 times the upper limits of normal) less than 6 months before the study
3. Know allergy to pyridine-containing drugs
4. Neurologic, degenerative, or psychiatric disorders that would impair the patient's ability to complete the protocol
5. Any illness or abnormality that would jeopardize patient safety or interfere with the conduct of the study
6. Inability to discontinue excluded concomitant drug therapy
7. Were pregnant or lactating
8. Had received any other investigational drug less tan 30 days before the study
9. History of drug or alcohol abuse
10. Treatment with and anti-spasticity compound and could not maintain a stable daily dosage
11. Had received any drug known to cause significant major organ toxicity less tan 3 months before the study
12. Peripheral neuropathy
13. Treatment with corticosteroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Sensory Function | From baseline at 6 months after treatment
  This function will be examined using the ASIA International Standards for the Neurological and Functional Classification of Spinal Cord Injury. Sensory function will be evaluated and qualify for two modes, pin prick / light touch in all dermatomes. The first one will be measured with the sharp and blunt end of a safety pin and the last one will be evaluated with a cotton ball. A scale of 3 points (0- 2) will be used depending on whether the modality is normal (2), diminished (1) or absent (0). A score of 2 for each of the 28 key sensory points tested on each side of the body would result in a maximum score of 56 for pin prick, 56 for light touch, and a total of 112, higher values represent a better outcome.
Changes in Motor function | From baseline at 6 months after treatment
  Motor function will be examined using the ASIA International Standards for the Neurological and Functional Classification of Spinal Cord Injury. Muscle strength will be evaluated in each of the 20 key muscles, five in each limb, representing segments of the spinal cord C5 through T1 and L2 through S1, using a six-point rating scale (0-5). There is a maximum score of 25 for each extremity, totaling 50 for the upper limbs and 50 for the lower limbs. Changes in motor score (total range from 0 to 100, higher values represent a better outcome).
Changes in the functional assement of Spinal Cord Independence | From baseline at 6 months after treatment
  The Spinal Cord Independence Measure version III (SCIM III) has 16 questions on self-care, respiratory and sphincter management and mobility in and out of home, which ranges from 0 (total dependence) to 100 points (total Independence).
Changes in the Sphincters function | From baseline at 6 months after treatment
  The function of the anal sphincter and the bladder will be evaluated. The anal function will be qualified as a sensation when the patient can differentiate when the rectum is full and ready to empty and control when the patient can stop the fecal evacuation with enough time to reach the bathroom and eliminate the fecal material. The function of the bladder will be classified in the same way as the anal function. Positive or negative will be the final result of sensation and control.
Change of overall quality of life score as measured by Short Form-36 (SF-36) | From baseline at 6 months after treatment
  The Short Form-36 (SF-36) has 36 questions. Each question has a score, which will be transformed into a 0 to 100 scale, where 0 corresponds to "the worst health state" and 100 to "the best health state".
Changes in Mean International Index of Erectile Function | From baseline at 6 months after treatment
  The international Index of Erectile Function (IIEF) contains 15 questions, rated from 0 or 1 to 5, yielding an overall score of 5-75 points. A score of 1-10 indicates severe erectile dysfunction, 11-16 moderate dysfunction, 17-25 mild dysfunction, and greater than 25 "normal" function.
Incidence of Treatment-Emergent Adverse Events (Safety) | 6 months
  Safety will be measured by occurrence of Treatment-Emergent Adverse Events (TRAEs); data will represent the number of participants with abnormal laboratory values and/or adverse events that are related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Martín Paredes Cruz, MSc, Principal Investigator — Instituto Mexicano del Seguro Social; Israel Grijalva Otero, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de Especialidades, CMN Siglo XXI, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansebout RR, Blight AR, Fawcett S, Reddy K. 4-Aminopyridine in chronic spinal cord injury: a controlled, double-blind, crossover study in eight patients. J Neurotrauma. 1993 Spring;10(1):1-18. doi: 10.1089/neu.1993.10.1. PMID 8320728
- [Background] Waxman SG. Aminopyridines and the treatment of spinal cord injury. J Neurotrauma. 1993 Spring;10(1):19-24. doi: 10.1089/neu.1993.10.19. No abstract available. PMID 8320729
- [Background] Hayes KC, Blight AR, Potter PJ, Allatt RD, Hsieh JT, Wolfe DL, Lam S, Hamilton JT. Preclinical trial of 4-aminopyridine in patients with chronic spinal cord injury. Paraplegia. 1993 Apr;31(4):216-24. doi: 10.1038/sc.1993.40. PMID 8493036
- [Background] Hayes KC, Potter PJ, Wolfe DL, Hsieh JT, Delaney GA, Blight AR. 4-Aminopyridine-sensitive neurologic deficits in patients with spinal cord injury. J Neurotrauma. 1994 Aug;11(4):433-46. doi: 10.1089/neu.1994.11.433. PMID 7837283
- [Background] Zeidman SM, Ling GS, Ducker TB, Ellenbogen RG. Clinical applications of pharmacologic therapies for spinal cord injury. J Spinal Disord. 1996 Oct;9(5):367-80. PMID 8938604
- [Background] Potter PJ, Hayes KC, Hsieh JT, Delaney GA, Segal JL. Sustained improvements in neurological function in spinal cord injured patients treated with oral 4-aminopyridine: three cases. Spinal Cord. 1998 Mar;36(3):147-55. doi: 10.1038/sj.sc.3100559. PMID 9554012
- [Background] Hayes KC. 4-Aminopyridine and spinal cord injury: a review. Restor Neurol Neurosci. 1994 Jan 1;6(4):259-70. doi: 10.3233/RNN-1994-6401. PMID 21551756
- [Background] Donovan WH, Halter JA, Graves DE, Blight AR, Calvillo O, McCann MT, Sherwood AM, Castillo T, Parsons KC, Strayer JR. Intravenous infusion of 4-AP in chronic spinal cord injured subjects. Spinal Cord. 2000 Jan;38(1):7-15. doi: 10.1038/sj.sc.3100931. PMID 10762192
- [Background] van der Bruggen MA, Huisman HB, Beckerman H, Bertelsmann FW, Polman CH, Lankhorst GJ. Randomized trial of 4-aminopyridine in patients with chronic incomplete spinal cord injury. J Neurol. 2001 Aug;248(8):665-71. doi: 10.1007/s004150170111. PMID 11569894
- [Background] Wolfe DL, Hayes KC, Hsieh JT, Potter PJ. Effects of 4-aminopyridine on motor evoked potentials in patients with spinal cord injury: a double-blinded, placebo-controlled crossover trial. J Neurotrauma. 2001 Aug;18(8):757-71. doi: 10.1089/089771501316919120. PMID 11526982
- [Background] Grijalva I, Guizar-Sahagun G, Castaneda-Hernandez G, Mino D, Maldonado-Julian H, Vidal-Cantu G, Ibarra A, Serra O, Salgado-Ceballos H, Arenas-Hernandez R. Efficacy and safety of 4-aminopyridine in patients with long-term spinal cord injury: a randomized, double-blind, placebo-controlled trial. Pharmacotherapy. 2003 Jul;23(7):823-34. doi: 10.1592/phco.23.7.823.32731. PMID 12885095
- [Background] Hayes KC, Potter PJ, Hsieh JT, Katz MA, Blight AR, Cohen R. Pharmacokinetics and safety of multiple oral doses of sustained-release 4-aminopyridine (Fampridine-SR) in subjects with chronic, incomplete spinal cord injury. Arch Phys Med Rehabil. 2004 Jan;85(1):29-34. doi: 10.1016/s0003-9993(03)00651-8. PMID 14970964
- [Background] DeForge D, Nymark J, Lemaire E, Gardner S, Hunt M, Martel L, Curran D, Barbeau H. Effect of 4-aminopyridine on gait in ambulatory spinal cord injuries: a double-blind, placebo-controlled, crossover trial. Spinal Cord. 2004 Dec;42(12):674-85. doi: 10.1038/sj.sc.3101653. PMID 15356676
- [Background] Cardenas DD, Ditunno J, Graziani V, Jackson AB, Lammertse D, Potter P, Sipski M, Cohen R, Blight AR. Phase 2 trial of sustained-release fampridine in chronic spinal cord injury. Spinal Cord. 2007 Feb;45(2):158-68. doi: 10.1038/sj.sc.3101947. Epub 2006 Jun 13. PMID 16773037
- [Background] Grijalva I, Garcia-Perez A, Diaz J, Aguilar S, Mino D, Santiago-Rodriguez E, Guizar-Sahagun G, Castaneda-Hernandez G, Maldonado-Julian H, Madrazo I. High doses of 4-aminopyridine improve functionality in chronic complete spinal cord injury patients with MRI evidence of cord continuity. Arch Med Res. 2010 Oct;41(7):567-75. doi: 10.1016/j.arcmed.2010.10.001. PMID 21167397
- [Background] Cardenas DD, Ditunno JF, Graziani V, McLain AB, Lammertse DP, Potter PJ, Alexander MS, Cohen R, Blight AR. Two phase 3, multicenter, randomized, placebo-controlled clinical trials of fampridine-SR for treatment of spasticity in chronic spinal cord injury. Spinal Cord. 2014 Jan;52(1):70-6. doi: 10.1038/sc.2013.137. Epub 2013 Nov 12. PMID 24216616